CLINICAL TRIAL: NCT07355959
Title: Cross-over, Randomized, Open Label Study to Assess the Efficacy and Pressure Maintenance of MOBIDERM Autofit Versus Bandages in the Management of Breast Cancer Related Lymphedema (BCRL) in Night-time Maintenance Phase.
Brief Title: Clinical Study to Assess the Efficacy and Pressure Maintenance of MOBIDERM Autofit Versus Bandages in the Management of Breast Cancer Related Lymphedema (BCRL) in Night-time Maintenance Phase.
Acronym: MOBISCAN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thuasne (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EC55_MOBISCAN
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Limb Lymphoedema
Keywords: Lymphedema of upper limb; Compression garments; Lymphedema management

STUDY DESIGN:
Intervention Model Description: Cross-over, randomized, open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: (Other): Night-time MOBIDERM Autofit for the 1st month (1st phase) and self-bandages at night for the 2nd month (2nd phase).
  Interventions: Device: MOBIDERM Autofit Armsleeve; Device: Self-bandages
- Group 2: (Other): Self-bandages at night for the 1st month (1st phase) then Night-time MOBIDERM Autofit for the 2nd month (2nd phase).
  Interventions: Device: MOBIDERM Autofit Armsleeve; Device: Self-bandages

INTERVENTIONS:
Device: MOBIDERM Autofit Armsleeve — The MOBIDERM Autofit Armsleeve will be worn by the patients at night for one month.
Device: Self-bandages — Self-bandages will be worn by the patients at night for one month.

SUMMARY:
The aim of this cross-over, randomized study is to assess the efficacy and pressure maintenance of MOBIDERM Autofit versus bandages in the management of Breast Cancer Related Lymphedema (BCRL) in night-time maintenance phase.

DETAILED DESCRIPTION:
In order to optimize treatment of lymphedema efficacy, THUASNE developed the standard Auto-Adjustable Armsleeve using the MOBIDERM technology, named MOBIDERM Autofit.

The device has already been evaluated in several clinical studies as an adjuvant treatment to daily compressive garment during night-time maintenance phase in women with Breast cancer related lymphedema.

The possibility to use this category of devices during both phases of lymphedema treatment has been reinforced recently by studies that showed a similar reduction in lymphedema volume with wraps versus conventional multilayer bandages [Ochalek et al., 2023,Borman et al., 2021].

The global objective of the MOBISCAN study is to reinforce the efficacy of MOBIDERM Autofit garment by assessing its efficacy and pressure maintenance versus bandages in the management of upper limb Lymphedema in night-time maintenance phase.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Unilateral upper limb lymphedema of stage I, II or III according to the criteria defined by the International Society of Lymphology, following breast cancer
3. Patient in maintenance phase of lymphedema treatment
4. Affected arm that fits with one of the standard sizes of the Auto- Adjustable MOBIDERM Autofit provided.
5. Signed informed consent prior to any study-mandated procedure.

Exclusion Criteria:

1. Active cellulitis / Infectious dermo-hypodermatitis
2. Lymphedema associated with active cancer needing acute chemotherapy
3. Motor and sensitive neurological deficiency / psychiatric or addictive disorders
4. Patients for whom compression is contraindicated, such as untreated infections, skin irritation, thrombosis: presence of skin lesions on the sleeve placement
5. Pregnant or breastfeeding patient
6. Participation to any other clinical study which has an impact on the different endpoints
7. Vulnerable patient, adults being the object of a legal protective measure or enable to express their consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Volume excess variation | 2 months (Inclusion, first month and second month visit)
  The primary endpoint of this study is to compare the volume excess variation of the upper limb between both conditions: MOBIDERM Autofit and self-bandages after one month of treatment, using the SCANECA 3D scanner.

SECONDARY OUTCOMES:
Evolution of affected upper limb volume: | 2 months (Inclusion, first month and second month visit)
  Evolution of affected upper limb volume between baseline and 1 month of treatment with MOBIDERM Autofit and self-bandages in patients with upper limb lymphedema.
Device pressure: | 2 months (Inclusion, first month and second month visit)
  The level of pressure under the devices will be measured with Picopress during the 3 patient visits for each patient.
Evolution of hand lymphedema: | 2 months (Inclusion, first month and second month visit)
  The volume of the hand related to healthy and to affected upper limb will be measured at baseline and the volume of the hand related to affected upper limb after one month of treatment with MOBIDERM Autofit and bandages with a digital measure device and/or tape measurement to check and compare the absence of migration of lymphedema towards the hand between both conditions.
Comfort / Ease of use / satisfaction: | 2 month visit
  A self-questionnaire will be completed by the patient at the end of the study when the patient tested each of the devices and is able to compare comfort, ease of use and satisfaction.
  A qualitative follow-up interview will be proposed to a dozen of patients at the end of the study to obtain their feed-back about their study treatments (overall experience, benefits of self-management, experience when putting on, taking off and adjusting the device).
Compliance: | 2 months
  The patient will complete a diary during the study to report the compliance with each device at night (Wear/not wear, number of hours).
Patient's safety | 2 months
  The Number and type of serious and non-serious Adverse Device Effects (ADE) with a focus on the cutaneous ADE will be collected during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Lindemann, Physician, Principal Investigator — Ödemzentrum Bad Berleburg Klinik "Haus am Schloßpark" Hochstr. 7 D 57319 Bad Berleburg
Locations (1):
- Ödemzentrum Bad Berleburg Klinik, Bad Berleburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cancer Information Sytem. https://www.wcrf.org/cancer-trends/worldwide-cancer-data/ (September 2023, date last accessed).